CLINICAL TRIAL: NCT06053736
Title: 1-Week Dispensing Evaluation of REVIVE™ Toric Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ROC2-23-008
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Refractive Ametropia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- REVIVE™ Toric Soft Contact Lenses (Experimental)
  Interventions: Device: REVIVE Contact Lens

INTERVENTIONS:
Device: REVIVE Contact Lens — REVIVE Contact Lens

SUMMARY:
Experienced soft contact lens wearing subjects will be enrolled in this 1-week, post-market, bilateral, repeated measures, dispensing study. All subjects will be seen for a Screening/Dispensing Visit at which informed consent will be obtained and eligibility will be assessed. If subjects satisfy all eligibility criteria and none of the exclusion criteria, subjects will be fit and dispensed study lenses. If unsuccessful in the dispensed lenses, additional lenses may be trialed. Once vision and lens fit are determined to be acceptable, eligible subjects will wear study lenses in both eyes for at least 8 hours per day (with the exception of the follow-up visits where the lenses should be worn for a minimum of 2 hours), for approximately 1 week (7 days +/-3 days). Measurements will be taken at the insertion visit and at the 7-day follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years or older on the date the Informed Consent Form (ICF) is signed and have capacity to read, understand and provide written voluntary informed consent.
2. Have physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings.
3. Have no active ocular disease or allergic conjunctivitis.
4. Not be using any topical ocular medications.
5. Be willing and able to follow instructions.
6. Have signed a statement of informed consent

Exclusion Criteria:

1. Participating in a conflicting study in the opinion of the Investigator.
2. Considered by the Investigator to not be a suitable candidate for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Mean logMAR Visual Acuity at 6m | At one week follow up
  Mean logMAR Visual Acuity at 6m

CONTACTS AND LOCATIONS:
Locations (1):
- Bausch & Lomb, Incorporated, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No